CLINICAL TRIAL: NCT06302959
Title: Clock Proteins as a Prognostic Marker for Disease Progression
Brief Title: Clock Proteins as Prognostic Markers
Acronym: CLOCK-PM
Status: Terminated | Type: Observational
Why Stopped: Recruitment failure
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 36-232 ex 23/24
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- healthy controls: For healthy controls, participation in this study lasts only one day. The following samples will be collected at three time-points on the same day (4 am, 12 pm, 8 pm):
  Blood sampling: 80 mL citrated whole blood and 10 mL serum will be collected. Collection of spontaneous sputum: at least 5 ml of sputum are collected. Saliva collection: Saliva is also collected at all three time-points.
- mild-to-moderate asthma: For patients with mild-to-moderate asthma, participation in this study lasts only one day.
  The following samples will be collected at three time-points on the same day (4 am, 12 pm, 8 pm):
  Blood sampling: 80 mL citrated whole blood and 10 mL serum will be collected. Collection of spontaneous sputum: at least 5 ml of sputum are collected. Saliva collection: Saliva is also collected at all three time-points.
- severe eosinophilic asthma: Patients with severe eosinophilic asthma, will be monitored (i) before mepolizumab treatment, (ii) after 4 months of mepolizumab treatment, (iii) once they reach remission under mepolizumab treatment. Mepolizumab is already approved for the treatment of severe eosinophilic asthma and is not administered for study purposes but as a standard treatment.
  On the day of participation, the following samples will be collected at three time-points (4 am, 12 pm, 8 pm):
  Blood sampling: 80 mL citrated whole blood and 10 mL serum will be collected. Collection of spontaneous sputum: at least 5 ml of sputum are collected. Saliva collection: Saliva is also collected at all three time-points.

SUMMARY:
Asthma is a chronic inflammatory disease of the airways that follows a strong circadian rhythm: Signs of inflammation and symptoms worsen especially in the early morning hours. The molecular circadian clock, which is a complex machinery of transcriptional and translational feedback loops, seems to reflect the inflammatory environment of peripheral blood leukocytes. Therefore, in this observational study the investigators will monitor the molecular circadian clock in patients with severe eosinophilic asthma before and during mepolizumab treatment. Our major goal is to evaluate the potential of the molecular circadian clock to serve as a prognostic marker for disease progression, treatment response or remission in patients with severe eosinophilic asthma. The molecular circadian clock will be monitored in blood and sputum leukocytes from patients with severe eosinophilic asthma before mepolizumab treatment, after 4 month of mepolizumab therapy, and once they reach remission under mepolizumab treatment. Effects will be compared to healthy controls and patients with mild-moderate asthma without mepolizumab treatment.

DETAILED DESCRIPTION:
Asthma is a heterogenous disease usually characterized by chronic airway inflammation that follows a strong circadian rhythm: Signs of inflammation and symptoms worsen especially in the early morning hours. Sudden death due to severe asthma attacks also tends to occur more frequently at night. Circadian rhythms are autonomous, self-sustained oscillations in biologic processes that follow a 24h-cycle and are entrained to environmental cues, the most important being light. At the cellular level, the circadian oscillator originates from a transcriptional/translational feedback loop comprised of several transcription factors and nuclear receptors.

Preliminary results indicate that the molecular circadian clock reflects the inflammatory environment of peripheral blood leukocytes. Thus, monitoring the molecular circadian clock will contribute to our understanding of asthma pathogenesis and treatment response and serve as a sensitive prognostic marker for disease progression and remission.

The primary objective of this observational study is to evaluate the potential of the molecular circadian clock to serve as a prognostic marker for disease progression, treatment response or remission. Therefore, the investigators will characterize the expression and activation of the molecular circadian clock components on the protein (flow cytometry) and messenger ribonucleic acid (mRNA) (quantitative polymerase chain reaction, qPCR) level in peripheral blood and sputum leukocyte subsets of healthy subjects, patients with mild-to-moderate asthma, patients with severe eosinophilic asthma (i) before and (ii) after 4 months of mepolizumab treatment, as well as (iii) after reaching remission under mepolizumab treatment. Results will be correlated with exacerbation rates and lung function parameters. As a secondary objective, the investigators will elucidate how the molecular circadian clock is regulated by the inflammatory environment and if anti-asthmatic drugs or therapeutic application of synthetic clock ligands may reverse the dysbalanced clock in asthma patients. Further, the investigators will assess the correlation between the expression and activation of the molecular circadian clock and the inflammatory state of the patients. Therefore, results will be correlated with patient's symptoms, quality of life and cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the participant after being informed
* Age 18-65
* Both sexes (male:female ratio of 2:3)
* Mild-to-moderate asthma, severe eosinophilic asthma according to the "Global Initiative for Asthma" (GINA) guidelines and healthy controls

Exclusion Criteria:

* Respiratory tract infections during the last 2 months
* severe comorbidities
* oral corticosteroids during the last month
* Shift workers
* Subjects with sleep disorders and/or receiving sleep medication
* Pregnant or breast-feeding women
* Control subjects with atopy and/or allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mild-to-moderate or severe eosinophilic asthma and healthy controls will be recruited for this study. Three individual groups within an age-range of 18 to 65 years and a male:female ratio of 2:3 will be studied:
  1. 20 age and gender matched healthy controls (1 visit)
  2. 20 patients with mild-to-moderate asthma (1 visit)
  3. 20-60 patients with SEA
     * before mepolizumab treatment (visit 1)
     * under mepolizumab treatment for 4 months (visit 2)
     * after reaching remission under mepolizumab treatment (visit 3)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Correlation between clock expression, exacerbation rate and lung function. | Up to three time points within 23 months.
  Expression and activation data from the molecular circadian clock will be corelated with the number of exacerbations within the last year and lung function parameters of the subjects [mainly Forced expiratory volume 1 (FEV1) and FEV1/Forced vital capacity (FVC) ratio].

SECONDARY OUTCOMES:
Correlation between clock expression, symptoms and quality of life. | Up to three time points within 23 months.
  Expression and activation data from the molecular circadian clock will be correlated with self-reported symptoms and quality of life. Quality of life will be assessed and scored by using a standardized Asthma Quality of life Questionnaire (AQLQ(S)), a 32-item questionnaire used to assess the physical, occupational, emotional, and social qualities of adults aged 17 to 70 years with asthma. Items are scored by a 7-point Likert scale (7 = not impaired at all; 1 = severely impaired). Thus, the AQLQ(S) has a minimum value of 32 (severely impaired) and a maximum value of 224 (not impaired).

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Böhm, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham PS, Jackson C, Chakraborty A, Cain J, Durrington HJ, Blaikley JF. Circadian regulation of pulmonary disease: the importance of timing. Clin Sci (Lond). 2023 Jun 14;137(11):895-912. doi: 10.1042/CS20220061. PMID 37314017
- [Background] Durrington HJ, Farrow SN, Loudon AS, Ray DW. The circadian clock and asthma. Thorax. 2014 Jan;69(1):90-2. doi: 10.1136/thoraxjnl-2013-203482. Epub 2013 May 23. PMID 23704227
- [Background] Carter SJ, Durrington HJ, Gibbs JE, Blaikley J, Loudon AS, Ray DW, Sabroe I. A matter of time: study of circadian clocks and their role in inflammation. J Leukoc Biol. 2016 Apr;99(4):549-60. doi: 10.1189/jlb.3RU1015-451R. Epub 2016 Feb 8. PMID 26856993